CLINICAL TRIAL: NCT05535439
Title: Prospective Randomized Controlled Study Comparing the Diagnostic Yield and Specimen Adequacy of Flex 19 G EBUS-TBNA Needles and 22 G EBUS-FNB Device for the Evaluation of Mediastinal and Hilar Lymphadenopathy
Brief Title: Diagnostic Yield & Specimen Adequacy of Flex 19 G vs 22 G EBUS Needle - A Randomized Controlled Trial
Acronym: EBUS-TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Ajmal Khan, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EBUS RCT 2022
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Mediastinal Lymphadenopathy; Hilar Lymphadenopathy
Keywords: EBUS TBNA; 22 G FNB Device; 19 G Needle; Mediastinal Lymphadenopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Cytologist and Histopathologist evaluating Diagnostic Yield and Specimen Accuracy will be blinded for type of needle used to minimize the potential of bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 19 G EBUS-TBNA Needle (Experimental): Mediastinal or Hilar Lymphadenopathy will be sampled by using 19 G EBUS-TBNA Needle
  Interventions: Procedure: EBUS-TBNA using 22 G EBUS-FNB Device OR 19 G EBUS-FNA needle
- 22 G EBUS-FNB Device (Experimental): Mediastinal or Hilar Lymphadenopathy will be sampled by using 22 G EBUS-FNB Device
  Interventions: Procedure: EBUS-TBNA using 22 G EBUS-FNB Device OR 19 G EBUS-FNA needle

INTERVENTIONS:
Procedure: EBUS-TBNA using 22 G EBUS-FNB Device OR 19 G EBUS-FNA needle — Both arm will be interventional where mediastinal lymph nodes will be sampled by two typs of needle

SUMMARY:
Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is the minimally invasive diagnostic modality for the evaluation of mediastinal and hilar lymph nodes (LNs). Traditionally, EBUS-TBNA is performed using either 21 gauge (G) or 22 G needle with a major limitation of inadequate sample especially when histologic assessment of tissue architecture is necessary such as in lympho-proliferative disorders and granulomatous inflammation. Although the specimen obtained with larger bore 19 G needle has been shown to be superior in terms of more cellular material and ability to subclassify malignant disease, it has more bloody samples. Recently a novel 22 G fine needle biopsy device (EBUS-FNB) has been introduced for endobronchial use after an experience gained from gastroenterology endoscopic ultrasound reporting high yield for core biopsies. FNB device has a unique design with 3 symmetrical, fully formed, cutting heels with 3 angled points to provide acquisition of FNB specimen in the form of a core tissue which might improve the overall diagnostic yield. Herein, investigators will study the diagnostic yield and safety of the 22 G EBUS-FNB needle with 19 G EBUS needle in the evaluation of mediastinal and hilar lymphadenopathy.

DETAILED DESCRIPTION:
Assessment of mediastinal lymph nodes and masses is crucial to establish the etiological diagnosis as well as staging in patients with lung cancer. EBUS guided TBNA has emerged as rapid minimally invasive technique to visualize the lymph nodes beyond the tracheal or bronchial wall and real time sampling of the mediastinal and hilar lymph nodes. For the evaluation of mediastinal lymphadenopathy, EBUS-TBNA is superior to conventional TBNA and almost equivalent in diagnostic yield with mediastinoscopy. Traditionally, EBUS-TBNA is performed using either 21 G or 22 G needle limited by small sample volume especially when histologic assessment of tissue architecture is necessary such as in lympho-proliferative disorders, and granulomatous inflammation. Over the years, there is continued technical improvisation, but the diagnostic yield varies in different institutions attributable to factors like number of samples and needle passes per lymph node, size of the needle and rapid onsite evaluation. Fine needle aspiration (FNA) needles of various size (21 G to 25 G) improves procedural outcome by achieving specific diagnosis without invasive surgical technique but they are inherently limited by small size of the needle used to obtain the sample. Quite often, repeat or alternative procedures are required due to small samples to provide all the information needed for the comprehensive evaluation and management of the patient. Introduction of large bore needles and core biopsy needles has added further improvement in diagnostic dimensions providing adequate samples for diagnosis and ancillary studies. with fewer passes. Many institutions still have a EBUS TBNA as a predominant approach for mediastinal sampling but several recent studies support a possible role of gauge-up needles and core needle biopsy to improve the overall diagnostic approach. Besides these technical aspects, direct tissue examination by trained personnel at the procedure site to assess the sample adequacy (Rapid On-Site Evaluation, ROSE) is an additional ideal method to improve overall diagnostic yield. However, the utility of ROSE needs further evaluation as the newer large bore or core biopsy needles makes ROSE less necessary for ensuring adequacy during EBUS TBNA due to its high diagnostic yield.

Traditionally, a 22 G EBUS TBNA needle is utilized in majority of center due to better maneuverability and lymph node opposition during its insertion into the node with an inherent limitation of lower volume of sample. A systematic review of 33 studies involving 2698 patients of lung cancer showed pooled probability of obtaining a sufficient sample of 94.5% which was adequate for anaplastic lymphoma (ALK) and epidermal growth factor receptor (EGFR) mutation but there was an uncertainty regarding sample suitability for next generation sequencing. Subsequently, a 21 G needle was introduced to acquire more tissue in the form of core biopsy like material for molecular profiling. However, comparative studies showed conflicting results for specimen adequacy and diagnostic yield between the two (21 G vs 22 G) needle sizes. Although there was a high success rate of diagnosis with both needles, better characterization of non-malignant diseases and histologic preservation of malignant disease was evident with 21 G needles. To enable the core tissue sampling with flexibility of needle a new Pro-Core needle was developed. However, a recent pilot study evaluating the Echo Tip Pro-Core needle showed no additional benefits to specimen adequacy when compared with conventional needles. In a randomized study of sarcoid patients, Recent study showed no difference in the sensitivity, specimen adequacy, or safety of EBUS-TBNA when performed with the Pro-Core or the conventional needle. Continual development to yield better results, a gauge-up 19 G needle was introduced to address the challenges with diagnostic accuracy in lymphoma and sarcoidosis. The flexibility of the 19 G needle with larger tissue specimen for cytology and histology assessment addressed some of the technical limitation of earlier EBUS-TBNA with no complications. The performance of 19 G needle in comparison to 21 G or 22 G needle showed no difference in diagnostic yield in multiple studies. Although the specimen obtained with gauge-up needles like 19 G needle has been shown to be superior in terms of more cellular material and ability to subclassify malignant or granulomatous disease, its utility is limited by more bloody samples. These reports suggests, in a subset of conditions which requires tissue architectures for establishing the diagnosis, a larger bore needles may be more useful.

Considering, no statistically significant difference in diagnostic yield in studies comparing different needle size, a FNB devise through an EBUS procuring exclusive core tissue might be beneficial. Although, the benefits of a 22 G FNB device showing improved diagnostic yield with core tissue in patients with gastrointestinal diseases, there is limited data showing benefits of FNB devise used through EBUS for mediastinal lymphadenopathy. The first retrospective study of 100 patients using EBUS FNB reported core biopsy sample in 87% patients with diagnostic yield approaching 97%.. Herein, investigators intend to study the diagnostic yield and safety of the 22 G EBUS-FNB needle in comparison with 19 G EBUS-FNA needle in the evaluation of mediastinal and hilar lymphadenopathy. Investigators hypothesize that both needle will have a similar diagnostic yield due to the acquisition of a better and core tissue specimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Radiographic features of mediastinal or hilar adenopathy (>10 mm in any axis)

Exclusion Criteria:

1. Hypoxemic patient (SpO2 < 92% on fraction of inspired oxygen (FiO2) >0.3
2. Patients receiving anticoagulants or having known bleeding diathesis
3. Patients with poor cardiopulmonary reserve or marked hypoxemia at rest
4. Accessibility of more convenient site to establish the diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 1 Week
  Defined as the proportion of subjects with a diagnostic EBUS-TBNA specimen if It provided a definitive diagnosis such as malignancy, infection (Tubercular, Fungal), sarcoidosis.
  Or Diagnosed as Reactive Lymphoid Hyperplasia

SECONDARY OUTCOMES:
The proportion of subjects with adequate sample | 1 Week
  A sample is defined as adequate in the presence of any of the following
  1. Germinal center fragments (centroblasts, histiocytes)
  2. At least 100 lymphocytes per field (evaluated in at least five fields at × 100 magnification) with <2 groups of contaminating bronchial cells per field
  3. Definite diagnosis is established irrespective of the number of lymphocytes
  4. For molecular testing, a sample with as little as 20% of cancer cells may be adequate
Adverse Events | During or within 24 hours of the procedure
  endobronchial bleeding, pneumothorax, hypoxemia, mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Ajmal Khan, MD, DM, Principal Investigator — SGPGIMS
Locations (1):
- Department of Pulmonary Medicine, SGPGIMS, Lucknow, U P, India

IPD SHARING:
Plan to Share IPD: No
Final Excel Sheet with individual data duly completed